CLINICAL TRIAL: NCT02254278
Title: A Randomized Phase II Trial for Patients With p16 Positive, Non-Smoking Associated, Locoregionally Advanced Oropharyngeal Cancer
Brief Title: Reduced-Dose Intensity-Modulated Radiation Therapy With or Without Cisplatin in Treating Patients With Advanced Oropharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-HN002; NCI-2014-01279 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-HN002 (Other: NRG Oncology); NRG-HN002 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Stage III Oropharyngeal Squamous Cell Carcinoma; Stage IVA Oropharyngeal Squamous Cell Carcinoma; Stage IVB Oropharyngeal Squamous Cell Carcinoma; Stage IVC Oropharyngeal Squamous Cell Carcinoma; Tongue Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMRT 6 weeks + cisplatin (Experimental): IMRT 6 weeks with concurrent cisplatin
  Interventions: Drug: Cisplatin; Radiation: IMRT 6 weeks
- IMRT 5 weeks (Experimental): IMRT 5 weeks
  Interventions: Radiation: IMRT 5 weeks

INTERVENTIONS:
Drug: Cisplatin — 40 mg/m2 IV (intravenously) weekly for 6 weeks
  Arms: IMRT 6 weeks + cisplatin
Radiation: IMRT 6 weeks — Intensity-modulated radiation therapy (IMRT), 30 fractions over 6 weeks, 5 fractions per week, 2 Gray per fraction to total dose of 60 Gy
  Other Names: Intensity-Modulated Radiotherapy
  Arms: IMRT 6 weeks + cisplatin
Radiation: IMRT 5 weeks — Intensity-modulated radiation therapy (IMRT), 30 fractions over 5 weeks, 6 fractions per week, 2 Gray per fraction to total dose of 60 Gy
  Other Names: Intensity-Modulated Radiotherapy
  Arms: IMRT 5 weeks

SUMMARY:
This randomized phase II trial studies the side effects and how well modestly reduced-dose intensity-modulated radiation therapy (IMRT) with or without cisplatin works in treating patients with oropharyngeal cancer that has spread to other places in the body (advanced). Radiation therapy uses high energy x rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether IMRT is more effective with or without cisplatin in treating patients with oropharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

-To select the arm(s) achieving a 2-year progression-free survival rate of >= 85% without unacceptable swallowing toxicity at 1 year.

SECONDARY OBJECTIVES:

* To determine patterns of failure (locoregional relapse versus distant) and survival -(overall and progression-free) at 6 months and 2 years.
* To determine acute toxicity profiles at the end of radiation therapy and at 1 and 6 months.
* To determine late toxicity profiles at 1 and 2 years.
* To determine patient-reported swallowing outcomes at 6 months and 1 and 2 years.
* To determine the predictive value of 12-14 week, post-treatment fludeoxyglucose F 18 (FDG)-positron emission tomography (PET)/computed tomography (CT) for locoregional control and progression free survival (PFS) at 2 years.
* To determine the predictive value of blood and tissue biomarkers for disease outcomes at 2 years.
* To determine swallowing recovery per videofluoroscopy imaging at 2 years.

After completion of study treatment, patients are followed at 1 and 3 months then every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria

Step 1: Registration:

1. Pathologically (histologically or cytologically) proven diagnosis of squamous cell carcinoma (including the histological variants papillary squamous cell carcinoma and basaloid squamous cell carcinoma) of the oropharynx (tonsil, base of tongue, soft palate, or oropharyngeal walls); cytologic diagnosis from a cervical lymph node is sufficient in the presence of clinical evidence of a primary tumor in the oropharynx. Clinical evidence should be documented, may consist of palpation, imaging, or endoscopic evaluation, and should be sufficient to estimate the size of the primary (for T stage).
2. Patients must have clinically or radiographically evident measurable disease at the primary site or at nodal stations. Tonsillectomy or local excision of the primary without removal of nodal disease is permitted, as is excision removing gross nodal disease but with intact primary site. Limited neck dissections retrieving ≤ 4 nodes are permitted and considered as non-therapeutic nodal excisions.
3. Immunohistochemical staining for p16 must be performed on tissue, and this tissue must be submitted for central review. Fine needle aspiration (FNA) biopsy specimens may be used as the sole diagnostic tissue if formalin-fixed paraffin-embedded cell block material is available for p16 immunohistochemistry. FNA specimens prepared with adequate p16 testing in this manner are acceptable to submit for central review. If the p16 preparation is not adequate, additional specimens will be required to establish p16 status. Centers are encouraged to contact the pathology chairs for clarification.
4. Clinical stage T1-T2, N1-N2b or T3, N0-N2b (AJCC, 7th ed.) including no distant metastases based on the following diagnostic workup:

   * General history and physical examination within 56 days prior to registration;
   * Fiberoptic exam with laryngopharyngoscopy (mirror and/or fiberoptic and/or direct procedure) within 70 days prior to registration;
   * One of the following combinations of imaging is required within 56 days prior to registration:

     1. A computed tomography (CT) scan of the neck (with contrast) and a chest CT scan (with or without contrast);
     2. or an MRI of the neck (with contrast) and a chest CT scan (with or without contrast);
     3. or a CT scan of neck (with contrast) and a PET/CT of neck and chest (with or without contrast);
     4. or an MRI of the neck (with contrast) and a PET/CT of neck and chest (with or without contrast).

   Note: A CT scan of neck and/or a PET/CT performed for the purposes of radiation planning may serve as both staging and planning tools.
5. Patients must provide their personal smoking history prior to registration. The lifetime cumulative history cannot exceed 10 pack-years. The following formula is used to calculate the pack-years during the periods of smoking in the patient's life; the cumulative total of the number of pack-years during each period of active smoking is the lifetime cumulative history.

   Number of pack-years = [Frequency of smoking (number of cigarettes per day) × duration of cigarette smoking (years)] / 20

   Note: Twenty cigarettes is considered equivalent to one pack. The effect of non-cigarette tobacco products on the survival of patients with p16-positive oropharyngeal cancers is undefined. While there are reportedly increased risks of head and neck cancer associated with sustained heavy cigar and pipe use (Wyss 2013), such sustained use of non-cigarette products is unusual and does not appear to convey added risk with synchronous cigarette smoking. Cigar and pipe tobacco consumption is therefore not included in calculating the lifetime pack-years. Marijuana consumption is likewise not considered in this calculation. There is no clear scientific evidence regarding the role of chewing tobacco-containing products in this disease, although this is possibly more concerning given the proximity of the oral cavity and oropharynx. In any case, investigators are discouraged from enrolling patients with a history of very sustained use (such as several years or more) of non-cigarette tobacco products alone.
6. Zubrod Performance Status of 0-1 within 56 days prior to registration;
7. Age ≥ 18;
8. The trial is open to both genders;
9. Adequate hematologic function within 14 days prior to registration, defined as follows:

   * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3;
   * Platelets ≥ 100,000 cells/mm3;
   * Hemoglobin (Hgb) ≥ 8.0 g/dl; Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.
10. Adequate renal function within 14 days prior to registration, defined as follows:

    • Serum creatinine (Cr) < 1.5 mg/dl or creatinine clearance (CC) ≥ 50 ml/min determined by 24-hour collection or estimated by Cockcroft-Gault formula:
    * CC male = [(140 - age) x (wt in kg)] / [(Serum Cr mg/dl) x (72)]
    * CC female = 0.85 x (CC male)
11. Adequate hepatic function within 14 days prior to registration defined as follows:

    * Bilirubin < 2 mg/dl;
    * Aspartate transaminase (AST) or alanine transaminase (ALT) < 3 x the upper limit of normal.
12. Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential;
13. Patients who are HIV positive but have no prior Acquired Immune Deficiency Syndrome (AIDS) -defining illness and have CD4 cells of at least 350/mm3 are eligible. HIV-positive patients must not have multi-drug resistant HIV infection or other concurrent AIDS-defining conditions. Patients must not be sero-positive for Hepatitis B (Hepatitis B surface antigen positive or anti-hepatitis B core antigen positive) or sero-positive for Hepatitis C (anti-Hepatitis C antibody positive). However, patients who are immune to hepatitis B (anti-Hepatitis B surface antibody positive) are eligible (e.g. patients immunized against hepatitis B).
14. The patient must provide study-specific informed consent prior to study entry, including consent for mandatory submission of tissue for required, central p16 review.
15. Patients who speak English (or read one of the languages for which a translation is available (see Section 10.2) must consent to complete the mandatory dysphagia-related patient reported instrument (MDADI). If the patient cannot understand spoken English and reads only languages not available in the MDADI translations, the patient can still participate in the trial, as this has been factored into the trial statistics. For all other patients, the MDADI is mandatory as it is included in the primary endpoint to be studied.

    Step 2: Randomization:
16. p16 positive by immunohistochemistry (defined as greater than 70% strong nuclear or nuclear and cytoplasmic staining of tumor cells), confirmed by central pathology review; (see Section 10.1 for details).

Exclusion Criteria

Step 1: Registration:

1. Cancers considered to be from an oral cavity site (oral tongue, floor mouth, alveolar ridge, buccal or lip), or the nasopharynx, hypopharynx, or larynx, even if p16 positive, or histologies of adenosquamous, verrucous, or spindle cell carcinomas;
2. Carcinoma of the neck of unknown primary site origin (even if p16 positive);
3. Radiographically matted nodes, defined as 3 abutting nodes with loss of the intervening fat plane;
4. Supraclavicular nodes, defined as nodes visualized on the same axial imaging slice as the clavicle;
5. Definitive clinical or radiologic evidence of metastatic disease or adenopathy below the clavicles;
6. Gross total excision of both primary and nodal disease with curative intent; this includes tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease. In other words, to participate in this protocol, the patient must have clinically or radiographically evident gross disease for which disease response can be assessed.
7. Patients with simultaneous primary cancers or separate bilateral primary tumor sites are excluded with the exception of patients with bilateral tonsil cancers;
8. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1095 days (3 years) (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible);
9. Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable;
10. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
11. Severe, active co-morbidity defined as follows:

    * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
    * Transmural myocardial infarction within the last 6 months;
    * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
    * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration;
    * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol other than those requested in Section 3.2.10.
    * Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition with immune compromise greater than that noted in Inclusion Criterion 13; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
12. Pregnancy; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
13. Prior allergic reaction to cisplatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Yom, Principal Investigator — NRG Oncology
Locations (222):
- United States (207):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Marin General Hospital, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Yale University, New Haven, Connecticut
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Mission Hospital, Asheville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Tennessee Cancer Specialists-Dowell Springs, Knoxville, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (13):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Island Cancer Centre, Victoria, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Saint Lukes Hospital, Dublin, Co Dublin, Ireland
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Yom SS, Torres-Saavedra P, Caudell JJ, Waldron JN, Gillison ML, Xia P, Truong MT, Kong C, Jordan R, Subramaniam RM, Yao M, Chung CH, Geiger JL, Chan JW, O'Sullivan B, Blakaj DM, Mell LK, Thorstad WL, Jones CU, Banerjee RN, Lominska C, Le QT. Reduced-Dose Radiation Therapy for HPV-Associated Oropharyngeal Carcinoma (NRG Oncology HN002). J Clin Oncol. 2021 Mar 20;39(9):956-965. doi: 10.1200/JCO.20.03128. Epub 2021 Jan 28. PMID 33507809

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After first step registration and prior to randomization, patients were tested for p16. Only patients with p16-positive tumors continued on to randomization. In total, 316 patients were enrolled and 308 were randomized.
Period: Overall Study
Arm/Group | IMRT 6 Weeks + Cisplatin | IMRT 5 Weeks
Started | 158 | 150
Eligible | 157 | 149
Started Study Treatment (Randomized and eligible participants who started study treatment) | 152 | 147
Negative Post-treatment PET (Randomized and eligible with negative post-treatment positron emission tomography (PET) scan) | 58 | 57
Completed (Participants contributing data to results are considered to have completed the study) | 157 | 149
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | IMRT 6 Weeks + Cisplatin | IMRT 5 Weeks | Total
Number analyzed (Participants) | 157 | 149 | 306
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 | 28 | 14 | 42
  50 - 59 | 56 | 60 | 116
  60 - 69 | 46 | 55 | 101
  ≥ 70 | 27 | 20 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 133 | 124 | 257
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 143 | 130 | 273
  Unknown or Not Reported | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 151 | 130 | 281
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 12 | 16
Zubrod performance status [Count of Participants; unit: Participants]
  0: Asymptomatic | 132 | 113 | 245
  1: Symptomatic but completely ambulatory | 25 | 36 | 61
Smoking history (pack years) [Count of Participants; unit: Participants] — Smoking history as measured in pack-years, calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked.
  Participants
    0 | 112 | 101 | 213
    >0 - <5 | 26 | 32 | 58
    5 - 10 | 19 | 16 | 35
Primary tumor site [Count of Participants; unit: Participants]
  Oropharynx NOS (not otherwise specified) | 4 | 13 | 17
  Tonsillar fossa, tonsil | 83 | 78 | 161
  Base of tongue | 68 | 58 | 126
  Pharyngeal oropharynx | 1 | 0 | 1
  Posterior pharyngeal wall | 1 | 0 | 1
T stage, clinical [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 7th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T1 | 64 | 51 | 115
    T2 | 67 | 80 | 147
    T3 | 26 | 18 | 44
N stage, clinical [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 7th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. The higher the number after the N, the greater the involvement of regional lymph nodes.
  Participants
    N0 | 6 | 7 | 13
    N1 | 28 | 34 | 62
    N2a | 24 | 19 | 43
    N2b | 99 | 89 | 188
Radiation Therapy (RT) planning (as stratified) [Count of Participants; unit: Participants] — Radiation therapy plan included unilateral or bilateral radiation to the neck, as provided by the treating site at stratification.
  Participants
    Unilateral | 52 | 47 | 99
    Bilateral | 105 | 102 | 207
RT planning (per central review) [Count of Participants; unit: Participants] — Radiation therapy plan included unilateral or bilateral radiation to the neck, as provided by central review by the study radiation oncologist.
  Participants
    Unilateral | 16 | 21 | 37
    Bilateral | 136 | 125 | 261
    Unknown | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Alive Without Progression at Two Years (Progression-free Survival)
Description: Progression is defined as local, regional, or distant disease progression or death due to any cause. Percentage is estimated using the binomial distribution.
Time Frame: From randomization to 2 years
Population: Two-year data was available for 147/157 (Arm 1) and 145/149 (Arm 2) randomized and eligible participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- IMRT 6 Weeks + Cisplatin (Arm 1): Cisplatin: 40 mg/m2 IV (intravenously) weekly for 6 weeks
  IMRT 6 weeks: Intensity-modulated radiation therapy (IMRT), 30 fractions over 6 weeks, 5 fractions per week, 2 Gray per fraction to total dose of 60 Gy
- IMRT 5 Weeks (Arm 2): IMRT 5 weeks: Intensity-modulated radiation therapy (IMRT), 30 fractions over 5 weeks, 6 fractions per week, 2 Gray per fraction to total dose of 60 Gy
Arm/Group | IMRT 6 Weeks + Cisplatin (Arm 1) | IMRT 5 Weeks (Arm 2)
Number analyzed (Participants) | 147 | 145
percentage of participants | 90.5 [86.6 to NA] — one-side confidence interval | 87.6 [83.3 to NA] — one-side confidence interval
Statistical Analysis 1: Comparison: IMRT 6 Weeks + Cisplatin (Arm 1); Assuming a binomial distribution, 140 eligible patients per arm were required for 80% power and 1-sided type I error rate of 10% to test the null hypothesis of 2-year progression-free survival (PFS) rate ≤ 85% against the alternative hypothesis of > 85% with a binomial test. The arms are not compared to each other; they are each tested separately against the null hypothesis; Test type: Superiority; p = 0.04, binomial; One-sided significance level=0.10
Statistical Analysis 2: Comparison: IMRT 5 Weeks (Arm 2); Assuming a binomial distribution, 140 eligible patients per arm were required for 80% power and 1-sided type I error rate of 10% to test the null hypothesis of 2-year PFS rate ≤ 85% against the alternative hypothesis of > 85% with a binomial test. The arms are not compared to each other; they are each tested separately against the null hypothesis; Test type: Superiority; p = 0.23, bionmial; One-sided significance level = 0.10

2. Secondary Outcome: Percentage of Participants With Local-regional Failure
Description: Local-regional failure is defined as local or regional progression, salvage surgery of the primary tumor with tumor present/unknown, salvage neck dissection with tumor present/unknown > 20 weeks after the end of radiation therapy, death due to study cancer without documented progression, or death due to unknown causes without documented progression. Distant metastasis and death due to other causes are considered competing risks. Local-regional failure time is defined as time from randomization to the date of first progression/death or last known follow-up (censored). Rates are estimated by the cumulative incidence method.
Time Frame: From randomization to 2 years
Population: Randomized and eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT 6 Weeks + Cisplatin | IMRT 5 Weeks
Number analyzed (Participants) | 157 | 149
percentage of participants
  Six months | 0.7 [0.1 to 3.3] | 2.0 [0.6 to 5.4]
  Two years | 3.3 [1.2 to 7.1] | 9.5 [5.5 to 15.0]
Statistical Analysis 1: Comparison: IMRT 6 Weeks + Cisplatin vs IMRT 5 Weeks; Test type: Superiority; p = 0.02, Log Rank; Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.17 to 0.90] — Reference level = IMRT 5 weeks

3. Secondary Outcome: Percentage of Participants With Distant Metastasis
Description: Distant metastasis is defined as distant progression. Local-regional failure and death due to any cause are considered competing risks. Distant metastasis time is defined as time from randomization to the date of progression/death or last known follow-up (censored). Rates are estimated by the cumulative incidence method.
Time Frame: From randomization to 2 years
Population: Randomized and eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT 6 Weeks + Cisplatin | IMRT 5 Weeks
Number analyzed (Participants) | 157 | 149
percentage of participants
  Six months | 0 [0 to 0] | 0 [0 to 0]
  Two years | 4.0 [1.6 to 8.0] | 2.1 [0.6 to 5.5]
Statistical Analysis 1: Comparison: IMRT 6 Weeks + Cisplatin vs IMRT 5 Weeks; Test type: Superiority; p = 0.58, Log Rank; Two-sided significance level = 0.05; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.4 to 5.08] — Reference level = IMRT 5 weeks

4. Secondary Outcome: Percentage of Participants Alive
Description: Overall survival time is defined as time from randomization to the date of death or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method.
Time Frame: from randomization to 2 years
Population: Randomized and eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT 6 Weeks + Cisplatin | IMRT 5 Weeks
Number analyzed (Participants) | 157 | 149
percentage of participants
  Six months | 99.3 [98.1 to 100] | 98.0 [95.7 to 100]
  Two years | 96.7 [93.9 to 99.5] | 97.3 [94.6 to 99.9]
Statistical Analysis 1: Comparison: IMRT 6 Weeks + Cisplatin vs IMRT 5 Weeks; Test type: Superiority; p = 0.93, Log Rank — Two-side significance level = 0.05; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.31 to 2.95] — Reference level = IMRT 5 weeks

5. Secondary Outcome: Percentage of Participants With Grade 3+ Adverse Events
Description: Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE.
Time Frame: End of radiation therapy (RT) (approximately 6 weeks for Arm 1 and 5 weeks for Arm 2), then 1 month, 6 months, 1 year, and two years after end of RT
Population: Randomized and eligible participants who started study treatment. Adverse event data was not available for all participants at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT 6 Weeks + Cisplatin (Arm 1) | IMRT 5 Weeks (Arm 2)
Number analyzed (Participants) | 152 | 147
percentage of participants
  End of RT | 73.7 [65.9 to 80.5] | 46.3 [38.0 to 54.7]
  1 month post-RT: number analyzed (Participants) | 144 | 142
  1 month post-RT | 36.1 [28.3 to 44.5] | 28.2 [21.0 to 36.3]
  6 months post-RT: number analyzed (Participants) | 140 | 126
  6 months post-RT | 17.9 [11.9 to 25.2] | 11.1 [6.2 to 17.9]
  1 year post-RT: number analyzed (Participants) | 143 | 134
  1 year post-RT | 14.0 [8.8 to 20.8] | 9.0 [4.7 to 15.1]
  2 years post-RT: number analyzed (Participants) | 128 | 122
  2 years post-RT | 8.6 [4.4 to 14.9] | 7.4 [3.4 to 13.5]
Statistical Analysis 1: Comparison: IMRT 6 Weeks + Cisplatin (Arm 1) vs IMRT 5 Weeks (Arm 2); End of RT; Test type: Superiority; p < 0.0001, Fisher Exact; Two-sided significance level = 0.05
Statistical Analysis 2: Comparison: IMRT 6 Weeks + Cisplatin (Arm 1) vs IMRT 5 Weeks (Arm 2); One month after end of RT; Test type: Superiority; p = 0.17, Fisher Exact; Two-sided significance level = 0.05
Statistical Analysis 3: Comparison: IMRT 6 Weeks + Cisplatin (Arm 1) vs IMRT 5 Weeks (Arm 2); Six months after end of RT; Test type: Superiority; p = 0.16, Fisher Exact; Two-side significance level = 0.05
Statistical Analysis 4: Comparison: IMRT 6 Weeks + Cisplatin (Arm 1) vs IMRT 5 Weeks (Arm 2); One year after end of RT; Test type: Superiority; p = 0.26, Fisher Exact; Two-side significance level = 0.05
Statistical Analysis 5: Comparison: IMRT 6 Weeks + Cisplatin (Arm 1) vs IMRT 5 Weeks (Arm 2); Two years after the end of RT; Test type: Superiority; p = 0.82, Fisher Exact; Two-side significance level = 0.05

6. Secondary Outcome: Mean One-year Total MD Anderson Dysphagia Inventory (MDADI) Score (Patient-reported Swallowing Outcome)
Description: The MDADI is a 20-item tool with each item scored as Strongly agree; Agree; No opinion; Disagree; or Strongly disagree. There is 1 global item (G1), 6 emotional subscale items (E2-E7), 5 functional subscale items (F1-F5), and 8 physical subscale items (P1-P8). For all items except E7 and F2, Strongly agree corresponds to a score of 1, Agree 2, No opinion 3, Disagree 4, and Strongly disagree 5. For E7 and F2, the scores are reversed; these 2 items are rescored to match the others before calculating summary scores. The composite (total) score is the mean of the 19 items (other than G1) X 20. Composite scores range from 20 to 100 with higher scores indicating less dysphagia.
Time Frame: One year post-RT. Radiation therapy (RT) ends at approximately 6 weeks for Arm 1 and 5 weeks for Arm 2
Population: Randomized and eligible participants. Questionnaires were not completed by all participants. 121 Arm 1 and 106 Arm 2 participants had one year post-RT data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | IMRT 6 Weeks + Cisplatin (Arm 1) | IMRT 5 Weeks (Arm 2)
Number analyzed (Participants) | 121 | 106
score on a scale | 85.3 [82.5 to 88.1] | 81.8 [79.0 to 84.5]

7. Secondary Outcome: Negative Predictive Value (NPV) of Post-treatment FDG-PET/CT Scan [Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET)/Computed Tomography (CT)] for Progression-free Survival and Local-regional Control at Two Years
Description: NPV is the percentage of participants alive and failure-free at 2 years among those with a negative post-treatment scan, as evaluated by central review. Negative scan determined as follows: primary site, right neck, left neck evaluated using a 5-point ordinal scale: 1-Definite complete metabolic response (CMR), 2-Likely CMR, 3-Likely inflammatory, 4-Likely residual metabolic disease (RMD), and 5-Definite RMD. 'Negative'= 1 or 2, 'Indeterminate'=3, 'Positive' = 4 or 5. 'Negative' for all three evaluation sites = overall score of 'Negative.' Progression (failure) is defined as local, regional, or distant disease progression (PR) or any death. Local-regional progression (failure) is defined as local or regional PR, salvage surgery of the primary tumor with tumor present/unknown, salvage neck dissection with tumor present/unknown > 20 weeks post RT, death due to study cancer or unknown causes without documented PR. The protocol specified that both arms would be combined for analysis.
Time Frame: 3 months (scan) and two years after the end of RT (approximately 6 weeks for Arm 1 and 5 weeks for Arm 2)
Population: Randomized and eligible participants with negative post-treatment PET
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Both Arms Combined: IMRT 6 Weeks + Cisplatin arm: Cisplatin: 40 mg/m2 IV (intravenously) weekly for 6 weeks; Intensity-modulated radiation therapy (IMRT), 30 fractions over 6 weeks, 5 fractions per week, 2 Gray per fraction to total dose of 60 Gy.
  IMRT 5 weeks arm: Intensity-modulated radiation therapy (IMRT), 30 fractions over 5 weeks, 6 fractions per week, 2 Gray per fraction to total dose of 60 Gy
Arm/Group | Both Arms Combined
Number analyzed (Participants) | 115
percentage of participants
  Progression-free Survival | 92.0 [87.7 to NA] — One-sided interval
  Local-regional failure | 94.5 [90.6 to NA] — One-side interval
Statistical Analysis 1: Comparison: Both Arms Combined; Progression-free survival: The null hypothesis of negative predictive value ≤ 90% was tested against the alternative of > 90% with a 1-sided binomial test at the 0.10 level; Test type: Superiority; p = 0.3, binomial test; One-sided significance level = 0.10
Statistical Analysis 2: Comparison: Both Arms Combined; Local-regional control: The null hypothesis of negative predictive value ≤ 90% was tested against the alternative of > 90% with a 1-sided binomial test at the 0.10 level; Test type: Superiority; p = 0.07, binomial test; One-sided significance level = 0.10

8. Secondary Outcome: Percentage of Participants Positive for Human Papillomavirus (HPV) Deoxyribonucleic Acid (DNA) After Treatment (Detection Rate)
Description: Positive HPV DNA status is defined as 5 or more HPV DNA fragments per mL of blood plasma, assessed by tumor-tissue modified viral (TTMV) testing.
Time Frame: Between 2 weeks to 1 month after treatment completion (approximately 6 weeks).
Population: Eligible participants with post-treatment HPV DNA value
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT 6 Weeks + Cisplatin (Arm 1) | IMRT 5 Weeks (Arm 2)
Number analyzed (Participants) | 60 | 69
percentage of participants | 3.3 [0.4 to 11.5] | 8.7 [3.3 to 18.0]
Statistical Analysis 1: Comparison: IMRT 6 Weeks + Cisplatin (Arm 1) vs IMRT 5 Weeks (Arm 2); Test type: Superiority; p = 0.28, Fisher Exact; Two-sided significance level = 0.05

9. Secondary Outcome: Change in Number of HPV DNA Fragments/mL (Copy Number) From Baseline to During Treatment (HPV DNA Rate Decline)
Description: Calculated as treatment value - baseline value. HPV DNA was assessed by tumor-tissue modified viral (TTMV) testing.
Time Frame: Baseline and during treatment (obtained after 20 Gy of radiotherapy and before 28 Gy, approximately between day 10 and 14)
Population: Eligible patients with baseline and during treatment HPV DNA values.
Measure: Mean (95% Confidence Interval); unit: fragments/mL
Arm/Group | IMRT 6 Weeks + Cisplatin (Arm 1) | IMRT 5 Weeks (Arm 2)
Number analyzed (Participants) | 70 | 69
fragments/mL | -1.06 [-1.68 to -0.45] | -0.22 [-0.68 to 0.24]
Statistical Analysis 1: Comparison: IMRT 6 Weeks + Cisplatin (Arm 1) vs IMRT 5 Weeks (Arm 2); Test type: Superiority; p = 0.03, t-test, 2 sided; Two-sided significance level = 0.05

10. Secondary Outcome: Correlation of Baseline Log HPV DNA Copy Number and Gross Tumor Volume (GTV)
Description: HPV DNA copy number is the number of HPV DNA fragments per mL of blood plasma, assessed by tumor-tissue modified viral (TTMV) testing. The natural logarithm of HPV DNA copy is used to determine correlation. GTV is the volume of the tumor determined by imaging used for treatment planning. The summary data of these two measures are reported separately in corresponding outcome measures. Correlation is measured by the Pearson correlation coefficient and ranges from -1 to +1, where ±1 indicates the strongest possible (negative or positive) correlation and 0 indicates no correlation. The study protocol indicates that participants are analyzed as a single group, treatment arms combined.
Time Frame: Baseline
Population: Eligible participants with baseline HPV DNA value
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Both Arms Combined
Number analyzed (Participants) | 164
correlation coefficient | 0.30 [0.15 to 0.44]

11. Secondary Outcome: Natural Logarithm (ln) of Baseline HPV DNA Copy Number [for Purpose of Correlation]
Description: HPV DNA copy number is the number of HPV DNA fragments per mL of blood plasma, assessed by tumor-tissue modified viral (TTMV) testing. The natural logarithm of HPV DNA copy is used to determine correlation with gross tumor volume. Note that a natural log, by definition, has no units. The study protocol indicates that participants are analyzed as a single group, treatment arms combined. Correlation of Baseline Log HPV DNA Copy Number and Gross Tumor Volume (GTV) are reported in another outcome measure.
Time Frame: Baseline
Population: Eligible participants with baseline HPV DNA value
Measure: Median (Full Range); unit: ln fragments per mL
Arm/Group | Both Arms Combined
Number analyzed (Participants) | 164
ln fragments per mL | 5.3 [0 to 12.2]

12. Secondary Outcome: Gross Tumor Volume (GTV) [for Purpose of Correlation]
Description: GTV is the volume of the tumor determined by imaging used for radiation treatment planning. The study protocol indicates that participants are analyzed as a single group, treatment arms combined. Correlation of Baseline Log HPV DNA Copy Number and Gross Tumor Volume (GTV) are reported in another outcome measure.
Time Frame: Baseline
Population: Eligible participants with baseline HPV DNA value
Measure: Median (Full Range); unit: mL
Arm/Group | Both Arms Combined
Number analyzed (Participants) | 164
mL | 25.7 [2.9 to 131.7]

13. Secondary Outcome: HPV DNA Status by 2-year Local-regional Failure Status
Description: Local-regional failure is defined as local or regional progression, salvage surgery of the primary tumor with tumor present/unknown, salvage neck dissection with tumor present/unknown > 20 weeks after the end of radiation therapy, death due to study cancer without documented progression, or death due to unknown causes without documented progression. Positive HPV DNA status is defined as 5 or more HPV DNA fragments per mL of blood plasma, assessed by tumor-tissue modified viral (TTMV) testing.
Time Frame: From end of treatment (approximate 6 weeks) to 2 years
Population: Eligible participants with post-treatment HPV DNA value and two-year local-regional failure data (i.e. not censored)
Measure: Count of Participants; unit: Participants
Groups:
- Local-regional Failure at 2 Years = No; Local-regional Failure at 2 Years = Yes: Treatment arms are combined:
  MRT 6 Weeks + Cisplatin arm: Cisplatin: 40 mg/m2 IV (intravenously) weekly for 6 weeks; Intensity-modulated radiation therapy (IMRT), 30 fractions over 6 weeks, 5 fractions per week, 2 Gray per fraction to total dose of 60 Gy.
  IMRT 5 weeks arm: Intensity-modulated radiation therapy (IMRT), 30 fractions over 5 weeks, 6 fractions per week, 2 Gray per fraction to total dose of 60 Gy
Arm/Group | Local-regional Failure at 2 Years = No | Local-regional Failure at 2 Years = Yes
Number analyzed (Participants) | 120 | 8
Participants
  HPV DNA Negative | 114 | 6
  HPV DNA Positive | 6 | 2
Statistical Analysis 1: Comparison: Local-regional Failure at 2 Years = No vs Local-regional Failure at 2 Years = Yes; Test type: Superiority; p = 0.08, Fisher Exact; Two-sided significance level = 0.05

14. Secondary Outcome: HPV DNA Status by 2-year Progression-free Survival Status
Description: Progression-free survival (PFS) failure is defined as local, regional, or distant disease progression or death due to any cause. Positive HPV DNA status is defined as 5 or more HPV DNA fragments per mL of blood plasma, assessed by tumor-tissue modified viral (TTMV) testing.
Time Frame: From end of treatment (approximate 6 weeks) to 2 years
Population: Eligible participants with post-treatment HPV DNA value and two-year progression-free survival data (i.e. not censored)
Measure: Count of Participants; unit: Participants
Groups:
- PFS Failure at 2 Years = No; PFS Failure at 2 Years = Yes: Treatment arms are combined:
  MRT 6 Weeks + Cisplatin arm: Cisplatin: 40 mg/m2 IV (intravenously) weekly for 6 weeks; Intensity-modulated radiation therapy (IMRT), 30 fractions over 6 weeks, 5 fractions per week, 2 Gray per fraction to total dose of 60 Gy.
  IMRT 5 weeks arm: Intensity-modulated radiation therapy (IMRT), 30 fractions over 5 weeks, 6 fractions per week, 2 Gray per fraction to total dose of 60 Gy
Arm/Group | PFS Failure at 2 Years = No | PFS Failure at 2 Years = Yes
Number analyzed (Participants) | 117 | 11
Participants
  HPV DNA Negative | 112 | 8
  HPV DNA Positive | 5 | 3
Statistical Analysis 1: Comparison: PFS Failure at 2 Years = No vs PFS Failure at 2 Years = Yes; Test type: Superiority; p = 0.02, Fisher Exact — Two-sided significance level = 0.05

ADVERSE EVENTS:
Time Frame: Weekly during treatment, at 1 and 3 months after end of treatment, then every 3 months from end of treatment for 2 years, every 6 months from end of treatment for 3 years, then annually until study completion. Maximum follow-up at time of reporting was 4.1 years.
Arm/Group | IMRT 6 Weeks + Cisplatin | IMRT 5 Weeks
All-Cause Mortality (participants affected / at risk) | 6/152 | 6/147
Serious Adverse Events (participants affected / at risk) | 31/152 | 11/147
Other Adverse Events (participants affected / at risk) | 152/152 | 147/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT 6 Weeks + Cisplatin (N=152) | IMRT 5 Weeks (N=147)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0
Heart failure (Cardiac disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 4 | 0
Esophagitis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 2 | 0
Flu like symptoms (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 1 | 0
Pain (General disorders) | 0 | 2
Appendicitis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Creatinine increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 6 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT 6 Weeks + Cisplatin (N=152) | IMRT 5 Weeks (N=147)
Anemia (Blood and lymphatic system disorders) | 92 | 35
Ear pain (Ear and labyrinth disorders) | 8 | 4
Hearing impaired (Ear and labyrinth disorders) | 43 | 34
Tinnitus (Ear and labyrinth disorders) | 65 | 41
Hypothyroidism (Endocrine disorders) | 18 | 16
Constipation (Gastrointestinal disorders) | 92 | 53
Diarrhea (Gastrointestinal disorders) | 26 | 14
Dry mouth (Gastrointestinal disorders) | 150 | 142
Dyspepsia (Gastrointestinal disorders) | 42 | 31
Dysphagia (Gastrointestinal disorders) | 124 | 119
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 | 3
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 16 | 13
Mucositis oral (Gastrointestinal disorders) | 131 | 121
Nausea (Gastrointestinal disorders) | 109 | 62
Oral pain (Gastrointestinal disorders) | 9 | 9
Vomiting (Gastrointestinal disorders) | 51 | 30
Fatigue (General disorders) | 138 | 117
Fever (General disorders) | 9 | 2
General disorders and administration site conditions - Other (General disorders) | 6 | 11
Neck edema (General disorders) | 4 | 10
Pain (General disorders) | 115 | 121
Infections and infestations - Other (Infections and infestations) | 12 | 7
Mucosal infection (Infections and infestations) | 10 | 10
Dermatitis radiation (Injury, poisoning and procedural complications) | 113 | 109
Alanine aminotransferase increased (Investigations) | 14 | 7
Aspartate aminotransferase increased (Investigations) | 12 | 7
Blood bilirubin increased (Investigations) | 9 | 5
Creatinine increased (Investigations) | 26 | 3
Lymphocyte count decreased (Investigations) | 118 | 87
Neutrophil count decreased (Investigations) | 33 | 3
Platelet count decreased (Investigations) | 53 | 8
Weight loss (Investigations) | 119 | 101
White blood cell decreased (Investigations) | 56 | 13
Anorexia (Metabolism and nutrition disorders) | 81 | 69
Dehydration (Metabolism and nutrition disorders) | 23 | 11
Hyperglycemia (Metabolism and nutrition disorders) | 27 | 13
Hyperkalemia (Metabolism and nutrition disorders) | 9 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 23 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 14 | 4
Hypokalemia (Metabolism and nutrition disorders) | 16 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 31 | 3
Hyponatremia (Metabolism and nutrition disorders) | 33 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 11
Trismus (Musculoskeletal and connective tissue disorders) | 22 | 25
Dizziness (Nervous system disorders) | 15 | 8
Dysgeusia (Nervous system disorders) | 142 | 132
Headache (Nervous system disorders) | 12 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 29 | 15
Anxiety (Psychiatric disorders) | 11 | 15
Depression (Psychiatric disorders) | 12 | 7
Insomnia (Psychiatric disorders) | 44 | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 37
Hiccups (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 18 | 19
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 29 | 44
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Sore throat (Respiratory, thoracic and mediastinal disorders) | 42 | 28
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 25
Dry skin (Skin and subcutaneous tissue disorders) | 36 | 35
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 12 | 10
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 9
Hypertension (Vascular disorders) | 10 | 11
Lymphedema (Vascular disorders) | 11 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT02254278/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT02254278/ICF_001.pdf